CLINICAL TRIAL: NCT02829983
Title: Clarithromycin as Adjuvant to Periodontal Debridement in the Treatment of Generalized Aggressive Periodontitis: Randomized Clinical Trial
Brief Title: Clarithromycin as Adjuvant to Periodontal Debridement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Estadual Paulista Júlio de Mesquita Filho (Other)
Collaborators: Coordenação de Aperfeiçoamento de Pessoal de Nível Superior. (Other Government)
Responsible Party: Principal Investigator, Mauro Pedrine Santamaria, DDS,MS,PhD, Universidade Estadual Paulista Júlio de Mesquita Filho
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: NMRBA
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Results first posted 2017-10-17 (Actual); Last update posted 2017-11-21 (Actual); Status verified 2017-10

CONDITIONS: Aggressive Periodontitis
Keywords: clarithromycin; periodontal debridement; aggressive periodontitis
MeSH Terms: conditions — Aggressive Periodontitis | interventions — Clarithromycin; Macrolides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- clarithromycin group (Active Comparator): 20 subjects that received one-stage full-mouth ultrasonic debridement (FMUD) associated with clarithromycin (500 mg - 12/12 hours) for 3 days.
  Interventions: Drug: Clarithromycin; Other: One-stage full-mouth ultrasonic debridement (FMUD)
- placebo group (Placebo Comparator): 20 subjects that received FMUD associated with placebo (members took with placebo 500 mg b.i.d. for 3 days).
  Interventions: Drug: Placebo; Other: One-stage full-mouth ultrasonic debridement (FMUD)

INTERVENTIONS:
Drug: Clarithromycin — Use of 500mg of Clarithromycin twice a day for 3 days
  Other Names: macrolide
  Arms: clarithromycin group
Drug: Placebo — Use of placebo tablets twice a day for 3 days.
  Arms: placebo group
Other: One-stage full-mouth ultrasonic debridement (FMUD) — One session of Periodontal debridement using ultrasonic device.

SUMMARY:
To assess the periodontal clinical response and the possible adverse effects of the clarithromycin combined to periodontal mechanical therapy in the treatment of patients with generalized aggressive periodontitis.

DETAILED DESCRIPTION:
To assess the periodontal clinical response and the possible adverse effects of the clarithromycin combined to periodontal mechanical therapy in the treatment of patients with generalized aggressive periodontitis.Forty patients were select and randomly assigned into two groups: Group clarithromycin with 20 subjects that received one-stage full-mouth ultrasonic debridement (FMUD) associated with clarithromycin (500 mg - 12/12 hours) for 3 days; group placebo with 20 subjects that received FMUD associated with placebo. Probing depth (PD), gain in clinical attachment level (CAL) and bleeding on probing (BOP) were evaluated at baseline, 3 and 6 months post- operatively.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of Generalized Aggressive Periodontitis
* presence of ≥20 teeth
* presence of ≥ 6 sites presenting probing depth (PD) ≥5mm with bleeding on probing (BOP) and ≥2 sites with PD ≥7mm (including incisors and first molars, in addition to two other non-contiguous teeth between them)
* good general health
* <35 years of age
* agree to participate in the study and sign a written consent

Exclusion Criteria:

* pregnant or lactating
* suffering from any other systemic disease (e.g. cardiovascular, diabetes, blood dyscrasias, immunodeficiency, etc) which could alter the course of periodontal disease
* received antimicrobials in the previous 6 months
* taking long-term anti-inflammatory drugs
* received a course of periodontal treatment within the last 12 months
* smoked

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2014-03; Primary Completion 2015-08 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mauro P Santamaria, DDS, PhD, Study Director — UPECLIN HC FM Botucatu Unesp

IPD SHARING:
Plan to Share IPD: Undecided
Undecided

REFERENCES:
- [Result] Casarin RC, Peloso Ribeiro ED, Sallum EA, Nociti FH Jr, Goncalves RB, Casati MZ. The combination of amoxicillin and metronidazole improves clinical and microbiologic results of one-stage, full-mouth, ultrasonic debridement in aggressive periodontitis treatment. J Periodontol. 2012 Aug;83(8):988-98. doi: 10.1902/jop.2012.110513. Epub 2012 Jan 30. PMID 22288485
- [Derived] Hammami C, Nasri W. Antibiotics in the Treatment of Periodontitis: A Systematic Review of the Literature. Int J Dent. 2021 Nov 8;2021:6846074. doi: 10.1155/2021/6846074. eCollection 2021. PMID 34790237
- [Derived] Khattri S, Kumbargere Nagraj S, Arora A, Eachempati P, Kusum CK, Bhat KG, Johnson TM, Lodi G. Adjunctive systemic antimicrobials for the non-surgical treatment of periodontitis. Cochrane Database Syst Rev. 2020 Nov 16;11(11):CD012568. doi: 10.1002/14651858.CD012568.pub2. PMID 33197289
- [Derived] Andere NMRB, Castro Dos Santos NC, Araujo CF, Mathias IF, Taiete T, Casarin RCV, Jardini MAN, Shaddox LM, Santamaria MP. Clarithromycin as an Adjunct to One-Stage Full-Mouth Ultrasonic Periodontal Debridement in Generalized Aggressive Periodontitis: A Randomized Controlled Clinical Trial. J Periodontol. 2017 Dec;88(12):1244-1252. doi: 10.1902/jop.2017.170165. Epub 2017 Jul 3. PMID 28671507

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Clarithromycin Group | Placebo Group
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Clarithromycin Group | Placebo Group | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 20 | 20 | 40
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 31.4 (3.7) | 31.25 (4.6) | 31.32 (0.10)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 19 | 38
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  Brazil | 20 | 20 | 40
Probing depht [Mean (Standard Deviation); unit: milimeter] | 3.34 (0.56) | 3.53 (0.6) | 3.43 (0.13)
clinical attachment level [Mean (Standard Deviation); unit: milimeter] | 3.48 (0.66) | 3.63 (0.7) | 3.55 (0.1)
bleeding on probing [Mean (Standard Deviation); unit: percentage of sites] | 53 (19) | 54 (30) | 53.5 (0.7)
gingival recession [Mean (Standard Deviation); unit: milimeter] | 0.14 (0.16) | 0.1 (0.12) | 0.12 (0.028)
plaque index [Mean (Standard Deviation); unit: percentage of sites] — Plaque index is the relation between the sites with deposits of plaque and the sites of full mouth divided for 100.
  percentage of sites | 59 (23) | 62 (25) | 60.5 (2.12)

OUTCOME MEASURES:

1. Primary Outcome: Clinical Attachment Level
Description: Distance from bottom of pocket to the cement-enamel junction (CEJ).
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: milimeter
Arm/Group | Clarithromycin Group | Placebo Group
Number analyzed (Participants) | 20 | 20
milimeter | 2.71 (0.35) | 3.03 (0.55)

2. Secondary Outcome: Probing Depth
Description: Distance from the bottom of sulcus/pocket to gingival margin
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: milimeter
Arm/Group | Clarithromycin Group | Placebo Group
Number analyzed (Participants) | 20 | 20
milimeter | 2.53 (0.3) | 2.86 (0.52)

ADVERSE EVENTS:
Time Frame: 1 week after periodontal treatment.
Arm/Group | Clarithromycin Group | Placebo Group
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 2/20 | 0/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Clarithromycin Group (N=20) | Placebo Group (N=20)
gastrointestinal discomfort (Gastrointestinal disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes